CLINICAL TRIAL: NCT06438653
Title: Reinterventions of Thoracic Endovascular Aortic Repair: a Retrospective Multicenter Cohort Study
Status: Active, not recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202312072RIND
Record Dates: First submitted 2024-05-27; First posted 2024-06-03 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-02

CONDITIONS: Thoracic Endovascular Aortic Repair
Keywords: Thoracic endovascular aortic repair; Reinterventions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Thoracic endovascular aortic repair
  Interventions: Other: No-intervenyion

INTERVENTIONS:
Other: No-intervenyion — No-intervenyion

SUMMARY:
We aimed to investigate the incidence of reinterventions in patients who underwent thoracic endovascular aortic repair (TEVAR) in multiple centers across Taiwan

DETAILED DESCRIPTION:
This study analyzed the multicenter data set for TEVAR procedures performed between 2012 and 2017. Each patient's survival was verified with a query to the national data set. Student's t-test and χ2 analysis were used to compare continuous and categorical variables between the groups that required reintervention and those that did not, respectively. Kaplan-Meier methods were applied to analyze freedom from reintervention and survival rates.We aimed to investigate the incidence of reinterventions in patients who underwent thoracic endovascular aortic repair (TEVAR) in multiple centers across Taiwan

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent thoracic endovascular aortic repair (TEVAR)

Exclusion Criteria:

* No thoracic endovascular aortic repair (TEVAR)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent thoracic endovascular aortic repair (TEVAR) in multiple centers across Taiwan.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Reintervention | 7 years
  The incidence of reinterventions in patients who underwent thoracic endovascular aortic repair (TEVAR)

SECONDARY OUTCOMES:
Mortality | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Yang Chan, phd, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes